CLINICAL TRIAL: NCT03213522
Title: A Comparison of Craniosacral Therapy vs Pelvic Floor Physical Therapy for the Treatment of Lower Urinary Tract Dysfunction in People With Multiple Sclerosis: A Pilot Study
Brief Title: Comparison of Craniosacral Therapy vs Pelvic Floor Physical Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CentraState Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CSMC 2016-14
Record Dates: First submitted 2017-04-17; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Multiple Sclerosis; Bladder Dysfunction; Urinary Incontinence; Overactive Bladder
MeSH Terms: conditions — Multiple Sclerosis; Urinary Incontinence; Urinary Bladder, Overactive | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic Floor Physical Therapy (Active Comparator): PFPT group will be treated/educated with/on therapeutic exercise, which includes, but not limited to, the pelvic brace, pelvic floor muscle exercise, and diaphragmatic breathing. If the patient is presenting with hypertonia of lower extremity muscles and/or muscles connecting to or part of the pelvic floor, the patient may be instructed on gentle static stretching and/or treated with passive stretching and diaphragmatic breathing.
  Interventions: Procedure: Pelvic Floor Physical Therapy
- CranioSacral Therapy (Active Comparator): Modified Upledger Institute 10-step protocol. Sequence of hand placements (for this protocol)/type of intervention which will mirror many of the treatment sequences described in the systematic review by Jakel and von Hauenschild (2012).
  Interventions: Procedure: Craniosacral Therapy

INTERVENTIONS:
Procedure: Pelvic Floor Physical Therapy — Educating the PFPT group on therapeutic exercise, which includes, but not limited to, the pelvic brace, pelvic floor muscle exercise, and diaphragmatic breathing. If the patient is presenting with hypertonia of lower extremity muscles and/or muscles connecting to or part of the pelvic floor, the patient may be instructed on gentle static stretching and/or treated with passive stretching and diaphragmatic breathing.
  Other Names: Bladder training; Pelvic floor muscle training; Prompted voiding
  Arms: Pelvic Floor Physical Therapy
Procedure: Craniosacral Therapy — Modified Upledger Institute 10-step protocol.
  Other Names: Osteopathic manipulation; Visceral manipulation
  Arms: CranioSacral Therapy

SUMMARY:
The purpose of this study is to determine the efficacy of CST for the treatment of LUTS in patients with MS and evaluate the acute effects compared to PFPT.

A. Objectives To examine the effect of CST as compared to PFPT on QOL, SEMG resting biofeedback readings, and PVR ultrasonography measures in patients with MS and LUTS.

B. Hypotheses / Research Question(s) It is hypothesized that patients who receive CST will demonstrate improved QOL, bladder control and ability to empty bladder as compared to those who receive PFPT.

DETAILED DESCRIPTION:
The purpose of this study is to determine if Craniosacral Therapy is an effective therapy for treating bladder dysfunction in patients with Multiple Sclerosis (MS). It will be compared to standard care for the treatment of bladder dysfunction, which is Pelvic Floor Physical Therapy. Bladder dysfunctions are extremely common in patients with Multiple Sclerosis. One of the most common symptoms of bladder dysfunction is called over-active bladder. Over- active bladder can be described by increased urges to urinate and frequency of urination, especially at night. Other common symptoms are: leakage of urine, with or without activity; inability to hold urine; and a decreased ability to empty bladder when urinating.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Multiple Sclerosis
* Currently have the following symptoms for at least three (3) months or longer: frequent urination, increased urge to urinate, nighttime urination, loss/leakage of urine with or without activity, and/or problems emptying your bladder.

Exclusion Criteria:

* Unable or unwilling to give consent to be treated
* Unable or unwilling to cover your portion of physical therapy treatment (i.e. co-pays and/or deductibles)
* Cannot speak or read English
* Have NOT had any urinary symptoms for at least three (3) months
* Do not have Multiple Sclerosis; or have NOT been diagnosed with Multiple Sclerosis
* Take medication to treat your urinary symptoms; or have taken medication in the past three (3) months to treat your urinary symptoms
* Use an indwelling catheter (i.e. tube inserted into your bladder for continuous urine drainage); or you require intermittent catheterization
* Currently are experiencing any of the following: shooting or radiating pain in your back or abdomen; pain that is not relieved with body position and/or medication; nausea; decreased appetite; pain with bowel movements or urination; and/or any symptom that is new and/or of unexplained onset (i.e. you do not know why it started or when it started)
* Currently have cancer/tumors (i.e. tumors in the spine, brain, pelvis, etc.) and/or aneurysms (i.e. abdominal aortic aneurysm)
* Received Botox injections in the past three (3) months
* Received Pelvic Floor Physical Therapy and/or Craniosacral Therapy in the past three (3) months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-04-10 (Actual); Primary Completion 2018-04-09 (Estimated); Study Completion 2018-04-09 (Estimated)

PRIMARY OUTCOMES:
PFDI-20 | Change from baseline PFDI-20 after six weeks of intervention
  Pelvic floor distress inventory self-report questionnaire
PFIQ-7 | Change from baseline PFIQ-7 after six weeks of intervention
  Pelvic floor incontinence questionnaire self-report

SECONDARY OUTCOMES:
MSQOL-54 | Change from baseline MSQOL-54 after six weeks of intervention
  Multiple Sclerosis Quality of Life self-report questionnaire
Post void residual volume | Change from baseline PVR after six weeks of intervention
  PVR measurement
Resting SEMG | Change from baseline Resting SEMG after six weeks of intervention
  surface electromyographic reading, resting only
Systolic BP | Change from baseline Systolic BP after six weeks of intervention
  blood pressure
Systolic BP | Change from pre-intervention to post-intervention at each of six intervention sessions
  blood pressure
Diastolic BP | Change from baseline Diastolic BP after six weeks of intervention
  blood pressure
Diastolic BP | Change from pre-intervention to post-intervention at each of six intervention sessions
  blood pressure
Pulse | Change from pre-intervention to post-intervention at each of six intervention sessions
  pulse
Pulse | Change from baseline Pulse after six weeks of intervention
  pulse

CONTACTS AND LOCATIONS:
Overall Officials: Danielle T Robbins, DPT, Principal Investigator — CentraState Medical Center
Locations (1):
- CentraState Medical Center, Freehold, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No